CLINICAL TRIAL: NCT00940030
Title: Effect of Mechanical Bowel Preparation With Polyethylene Glycol Plus Bowel Enema (Glycerine 5%) vs Bowel Enema Alone in Patients Candidates to Colorectal Resection for Malignancy. Prospective, Randomized Clinical Trial
Brief Title: Comparison of Mechanical Bowel Preparation Versus Enema for Candidates to Colorectal Resection for Adenocarcinoma
Acronym: MBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEO S357/307
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: Mechanical Bowel Preparation (MBP); enema
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Enema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBP+enema (Experimental): mechanical bowel preparation and enema
  Interventions: Other: mechanical bowel preparation; Other: enema
- enema (Active Comparator)
  Interventions: Other: enema

INTERVENTIONS:
Other: mechanical bowel preparation — fiberless diet starting 2 days before surgery. Drugs containing iron and coal plant will be stopped. Free breakfast the day before surgery. Lunch: meat broth and white meat. From 16 p. m. to 20 p. m. assumption of Polyethylene Glycol Macrogol 70 mg per 1 liter of water 4 times (1L each hour). A bowel enema (2L, glycerin 5%) will be administered at 6 a. m. the day of surgery.
  Arms: MBP+enema
Other: enema — fiberless diet starting 2 days before surgery. Drugs containing iron and coal plant will be stopped. Free breakfast the day before surgery. Lunch: meat broth and white meat. Dinner: meat broth and fasting starting from midnight. A bowel single enema (2L, glycerin 5%) will be administered at 6 a. m. the day of surgery.

SUMMARY:
The purpose of this study is to evaluate mechanical bowel preparation (MBP) with polyethylene glycol plus bowel enema versus bowel enema alone in patients candidates to colorectal resection for malignancy.

DETAILED DESCRIPTION:
Surgical site infections (SSI) in colorectal surgery (anastomotic leakage, wound infection, intraabdominal abscess) are associated with increased mortality, postoperative hospital stay and costs. From a recent metanalysis and randomized clinical trial there is the emerging evidence that mechanical bowel preparation (MBP) before elective colorectal surgery is not associated with reduction of SIS, although it causes high discomfort for patients. On the same way other more recent studies show that MBP may cause an higher incidence of SIS, and that MBP may alter the bowel mucosa morphology. Other Authors report an increased incidence of anastomotic leakage requiring surgery for patients undergoing a single preoperative phosphate enema whereas but an higher cardiovascular mortality for patients undergoing MBP. Two recent studies do not clarify the usefulness of MBP for reducing SIS after colorectal surgery and one stage anastomosis. For these reasons a more precise understanding of the relationship between MBP and SIS could increase patients satisfaction and decrease unnecessary procedures and costs. At this point MBP represent the clinical standard for patients undergoing elective colorectal surgery at the European Institute of Oncology.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates to colorectal surgery for histologically confirmed colorectal cancer
* Age 18-80 years
* Obtained written consent

Exclusion Criteria:

* Patients at high risk for receiving a stoma (e. g. patients affected by distal rectal cancer <5cm from the anal verge; patients whose tumour is located >5 cm from the anal verge who underwent neoadjuvant CT-RT without downstaging or tumour shrinkage
* Intestinal obstruction
* Emergency procedures
* Patients who underwent colonoscopy within 7 day from surgery
* ASA 4-5 patients
* Patients unable to give informed consent
* Renal failure (serum creatinine >3 mg/dl)
* Pregnant women
* Breast feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2007-10; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Anastomotic leakage, wound infection (including deep abscess) | 30 days after surgery

SECONDARY OUTCOMES:
post surgery extra abdominal complications | 30 days
patient's symptoms (through questionaire) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Andreoni, MD, Principal Investigator — European Institute of Oncology; Roberto Biffi, MD, Principal Investigator — European Institute of Oncology; Emilio Bertani, MD, Principal Investigator — European Institute of Oncolgy
Locations (1):
- European Institute of Oncology, Milan, Italy